CLINICAL TRIAL: NCT04755127
Title: ARthroscopiC SynovecTomy Versus Intra-Articular Injection of Corticosteroids for the Management of Therapy Refractory Psoriatic or Rheumatoid Arthritis of the Wrist: a Randomized Controlled Trial
Brief Title: Arthroscopic Synovectomy of the Wrist in Inflammatory Arthritis
Acronym: ARCTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maasstad Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARCTIC01
Record Dates: First submitted 2021-01-27; First posted 2021-02-15 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Wrist Arthritis; Psoriatic Arthritis; Rheumatoid Arthritis; Surgery
Keywords: Wrist arthroscopy; Arthroscopic synovectomy; Rheumatoid arthritis; Psoriatic Arthritis; Patient related outcome
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis, Rheumatoid | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: non-blinded randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular corticosteroid injection (Active Comparator): Injection with 40mg triamcinolone acetonide (kenacort) in the wrist
  Interventions: Drug: Intra-articular corticosteroid injection
- arthroscopic synovectomy (Experimental): Wrist arthroscopy in day surgery setting with debulking of synovitis, inspection of cartilage, ligament, tendon and bone damage, collection of synovial biopsies and deposition of intra-articular corticosteroids (40mg triamcinolone acetonide)
  Interventions: Procedure: Arthroscopic synovectomy of the wrist

INTERVENTIONS:
Procedure: Arthroscopic synovectomy of the wrist — Wrist arthroscopy in day surgery setting with debulking of synovitis, inspection of cartilage, ligament, tendon and bone damage, collection of synovial biopsies and deposition of intra-articular corticosteroids (40mg triamcinolone acetonide)
  Arms: arthroscopic synovectomy
Drug: Intra-articular corticosteroid injection — Injection with 40mg triamcinolone acetonide (kenacort) in the wrist
  Arms: Intra-articular corticosteroid injection

SUMMARY:
Rationale: Psoriatic (PsA) and rheumatoid arthritis (RA) are inflammatory joint diseases that often involve the wrist and may result in progressive joint destruction followed by impaired wrist function and reduced quality of life. The first line treatment usually consists of conventional Disease-Modifying Anti-Rheumatic Drugs (cDMARDs) along with bridging therapy using systemic corticosteroids or intra-articular corticosteroids in case of limited joint disease. After initiation therapy, intra-articular corticosteroids are often utilized as they provide rapid dampening of joint inflammation in case of a flare-up of disease activity (mono- or oligoarthritis). However, a substantial part of these patients clinically respond poorly or not at all. Alternatively, arthroscopic synovectomy may provide substantial relieve of symptoms, improve functionality, slow down disease progression and prevent joint destruction, as earlier studies have suggested. Prospective randomized studies are needed to confirm these findings. Moreover, they may prevent the need for expensive biological Disease-Modifying Anti-Rheumatic Drugs (bDMARDs) and assist in guiding therapeutic strategies in the long run, through collecting and analysing valuable synovial biopsies. Wrist arthroscopy is a routine procedure in the participating centres with only minor complications and fast recovery.

Objective: To compare arthroscopic synovectomy with deposition of intra-articular corticosteroids (DIACS) versus intra-articular injection of corticosteroids (IACSI) in RA and PsA patients with mono- or oligoarthritis of the wrist that is refractory to cDMARD therapy.

Study design: Multi-centre randomized controlled trial conducted in the Maasstad Hospital and Spijkenisse Medisch Centrum (SMC).

Study population: Patients with active RA or PsA and bDMARD-naive, who develop a localized flare of disease activity (mono- or oligoarthritis) that involves the wrist, defined as an increase in DAS28 > 1.2 or > 0.6 if DAS28 ≥ 3.2 compared to the last DAS28 measurement (maximum six months before) and that is refractory to systemic cDMARD for at least three months, defined as no response on the European League Against Rheumatism (EULAR) response criteria.

Intervention: This study will randomize between IACSI of the wrist (control) and arthroscopic synovectomy of the wrist combined with DIACS (intervention). During arthroscopy synovial biopsies will be collected and stored for later analysis of the functional and histological characteristics of the synovium (beyond the scope of this study).

Main study parameters/endpoints: Primary outcome is the change in Patient-Rated Wrist Evaluation (PRWE) score from randomization to three months of follow-up. The PRWE is a validated, fifteen-item self-reported questionnaire rating wrist pain and function. Secondary outcomes are resolution of wrist arthritis measured by ultrasound, standard wrist radiographs, DAS28, EULAR response rate, Visual Analogue Scale (VAS), EQ-5D quality of life questionnaire, iMTA Productivity Cost Questionnaire (iPCQ), iMTA Medical Consumption Questionnaire (iMCQ), cost effectiveness analyses (CEA), physical examination, adverse events (AE) and laboratory results. Follow-up visits are scheduled at three, six and twelve months after intervention.

Nature and extent of the burden and risks associated with study participation:

Both study arms include standard treatment of care. Wrist arthroscopy is a standard treatment for wrist arthritis and often implemented for other intra-articular wrist pathology. The risks include infection, neurovascular damage and articular surface damage. Nevertheless, wrist arthroscopy is a well-established and safe technique. Reduction of risks will be done according to inclusion and exclusion criteria. If complications arise, the treating physician will proportionate the adequate treatment according to the current protocols based on the published literature. Patients will be asked to return at three, six and twelve months. These visits are standard of care following the rheumatic arthritis protocol. Patients will be asked to complete questionnaires at baseline and at three follow-up moments. These will take 160 minutes in total. The arthroscopy group will return between ten to fourteen days for wound inspection. All patient will be contacted by telephone at two, four and six weeks for VAS pain scores.

Expected results: We expect that arthroscopic synovectomy followed by DIACS will lead to significantly more improvement in PRWE scores compared to IACSI three months after intervention. Furthermore, we anticipate that wrist arthroscopy will result in lower pain scores, better joint mobility, better response on EULAR score, sustained resolution of arthritis on ultrasound, less joint damage on radiographs and is more cost-effective after one-year analysis.

ELIGIBILITY:
Inclusion criteria In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Male and female patients with age ≥ 18 years
* Subjects able and willing to give written informed consent (or legally acceptable representative or impartial witness when applicable) and is available for entire study
* Patients meet the criteria of either group below:

Group 1. Inclusion criteria RA patients:

* Patients that are diagnosed with RA according to the revised 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Rheumatoid Arthritis Classification Criteria (table 1)
* Patients are experiencing an exacerbation defined as an increase in DAS28 > 1.2 or > 0.6 if DAS28 ≥ 3.2 compared to last DAS28 measurement (maximum six months before)
* The exacerbation is refractory to systemic cDMARDs for at least three months, defined as 'no response' according to the EULAR response criteria (table 2)
* Wrist arthritis, that is diagnosed clinically, is the predominant symptom

Group 2. Inclusion criteria PsA patients:

* Patients that are diagnosed with PsA according to the Classification Criteria for Psoriatic Arthritis (CASPAR) criteria (table 3)
* Patients are experiencing an exacerbation defined as an increase in DAS28 > 1.2 or > 0.6 if DAS28 ≥ 3.2 compared to last DAS28 measurement (maximum six months before)
* The exacerbation is refractory to systemic cDMARDs for at least three months, defined as 'no response' according to the EULAR response criteria (table 2)
* Wrist arthritis, that is diagnosed clinically, is the predominant symptom

Exclusion criteria A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Previous or current treatment with biological (b) DMARDs
* Current inflammatory joint disease other than RA or PsA (e.g. gout, reactive arthritis, Lyme disease)
* Subjects who are pregnant or intend to become pregnant during the study
* Intra-articular corticosteroids injection in the wrist in the last 6 months
* Previous wrist surgery
* Severe osteoarthritis with malformations of the wrist
* Congenital abnormalities of wrist function or motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Wrist evaluation (PRWE) | 3 months
  15-item questionnaire scoring pain and wrist function on a scale from 0-100, with a higher score indicating worse outcome.

SECONDARY OUTCOMES:
Patient-Rated Wrist evaluation (PRWE) | 6 and 12 months
  15-item questionnaire scoring pain and wrist function on a scale from 0-100, with a higher score indicating worse outcome.
Wrist ultrasound | 3 months
  Resolution of ultrasound (US) arthritis as defined by grey scale (B-mode) and power Doppler after three months compared to baseline measurement. Grey scale uses a two-dimensional image to visualize structural changes like synovial hypertrophy and bone erosions. Power Doppler mode can assess joint inflammatory activity by detecting pathological synovial blood flow. The EULAR-OMERACT (Outcome Measures in Rheumatology Clinical Trials) combined scoring system includes both greyscale and power Doppler and will be used to score arthritis in this study. Ultrasound has demonstrated greater sensitivity than clinical assessment and conventional radiography for detecting synovitis in RA target joints. Also, US signs of synovitis were found predictive for flare and failure of DMARD therapy, despite clinical remission. Furthermore, ultrasound techniques are low-invasive, inexpensive and require no radiation.
Wrist X-ray | 12 months
  Standard (plain) radiographs of the wrist at baseline and after twelve months. Arthritis on radiographs will be graded using the Modified Larsen grading system. This system grades wrist arthritis on a score of 0 to 5, 5 indicating the most joint abnormalities.
NRS pain score | 2, 4 and 6 weeks, 3, 6 and 12 months
  Numeric Rating Scale (NRS) pain score at baseline two, four and six weeks (by phone), and at three, six and twelve months (digitally). A score of 0 implies no pain and 10 the worst possible pain.
Range of motion | 3, 6 and 12 months
  Range of motion (ROM) of the wrist at baseline, three, six and twelve months. ROM will be measured actively with a goniometer and includes pronation, supination, ulnar and radial deviation and palmar and dorsal flexion.
Grip strength | 3, 6 and 12 months
  Grip strength of the wrist at baseline, three, six and twelve months. Grip strength will be measured using a dynamometer as the mean of three measurements.
DAS 28 | 3, 6 and 12 months
  EULAR response rate and Disease Activity Score (DAS28) at baseline, three, six and twelve months. The DAS28 is a measure of disease activity in rheumatoid arthritis in which 28 joints are examined for swelling and tenderness, combined with global pain scores and blood markers (www.DAS28-score.nl). The EULAR response rate measures responsiveness to anti-rheumatic treatment and is derived from the DAS28 score
EQ-5D | 3, 6 and 12 months
  EuroQol 5D (EQ-5D) at baseline, three, six and twelve months. The EQ-5D is a standardized questionnaire scoring quality of life on five different levels, on a scale from 0-100.
iPCQ questionnaire | 3, 6 and 12 months
  Institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (iPCQ) at baseline, three, six and twelve months. The iPCQ is a standardized instrument for measuring and valuing health related productivity losses. This wil be used for the cost effectiveness analysis.
iMCQ questionnaire | 3, 6 and 12 months
  Institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ) at baseline, three, six and twelve months. The iMCQ is a standardized instrument for measuring medical costs. The iMCQ includes questions related to frequently occurring contacts with health care providers, medication use and home care. This wil be used for the cost effectiveness analysis.
ESR | 3, 6 and 12 months
  Laboratory test: erythrocyte sedimentation rate (ESR) at baseline and three, six and twelve months (part of the routine clinical care).
CRP | 3, 6 and 12 months
  Laboratory tests: C-reactive protein (CRP) at baseline and three, six and twelve months (part of the routine clinical care).
Adverse events | One year
  Adverse events (AEs) (including glucocorticoid related AEs), AEs leading to withdrawal, AEs leading to discontinuation of medication, and AEs due to infusion reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Radjesh Bisoendial, MD, PhD, Principal Investigator — Maasstad ziekenhuis
Locations (1):
- Maasstad Hospital, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided